CLINICAL TRIAL: NCT00697281
Title: A Dose Finding Study Of The Effects Of OC000459 On Responses To Allergen Challenge In The Vienna Chamber In Subjects Known To Suffer From Grass Pollen Induced Allergic Rhinitis.
Brief Title: OC000459 Dose Finding Study in Hay Fever Sufferers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxagen Ltd (Industry)
Responsible Party: Dr C Mike Perkins, Oxagen Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OC000459/010/07
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; human; clinical trial; efficacy; safety; challenge test
MeSH Terms: conditions — Rhinitis, Allergic | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Dose level 1
  Interventions: Drug: OC000459
- 2 (Experimental): Dose level 2
  Interventions: Drug: OC000459
- 3 (Experimental): Dose level 3
  Interventions: Drug: OC000459
- 4 (Experimental): Dose level 4
  Interventions: Drug: OC000459
- 5 (Experimental): Dose level 5
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OC000459 — Tablets twice daily for 8 days
  Dose level 1
  Arms: 1
Drug: OC000459 — Tablets twice daily for 8 days
  Dose level 2
  Arms: 2
Drug: OC000459 — Tablets twice daily for 8 days
  Dose level 3
  Arms: 3
Drug: OC000459 — Tablets twice daily for 8 days
  Dose level 4
  Arms: 4
Drug: Placebo — Tablets twice daily for 8 days
  Dose level 5
  Arms: 5

SUMMARY:
The primary objective of this study is to evaluate a range of dose levels for efficacy in the control of symptoms of allergic rhinitis

DETAILED DESCRIPTION:
This will be a randomised, double blind, placebo controlled, parallel group evaluation of OC000459 given orally for eight days. Four dose levels will be studied and compared to placebo. They will be studied in treatment groups of 18 to 21 subjects. The placebo group will also consist of 18 to 21 subjects. There will be a screening period of up to six weeks. There will be a follow up one to three weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 50 years with a history of symptoms of grass pollen related allergic rhinitis within the previous two years.
* Females of childbearing potential (i.e. having had a menstrual period within two years prior to the date of screening) must practise two forms of contraception and must have a negative pregnancy test (blood or urine) at screening.
* Acceptable contraception includes the use of TWO of the following:

  * oral contraception (i.e. the Pill);
  * intrauterine device (an IUD or 'Coil');
  * barrier contraception (i.e. condoms or diaphragm/cap);
  * transdermal patch

Exclusion Criteria:

* Medical conditions likely to affect the outcome of the study.
* Nasal conditions likely to affect the outcome of the study, i.e. nasal septal perforations, nasal polyps, sinus disease, chronic nasal obstruction, or other nasal diseases as determined by the principal investigator or designee.
* Presence of any respiratory disease other than a history of mild stable asthma not requiring treatment and associated with normal lung function (defined as FEV1 ≥ 90% predicted for height and age).
* Immunotherapy treatment course in the past 28 days
* Use of inhaled or local corticosteroids in the past 28 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom score (TNSS) | After 8 days of treatment

SECONDARY OUTCOMES:
Other symptom scores of allergic rhinitis | After 8 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Univ Prof. Dr. Friedrich Horak, MD, Principal Investigator — Allergie Zentrum Wien West
Locations (1):
- Allergie Zentrum Wien West, Vienna Challenge Chamber, Vienna, Austria